CLINICAL TRIAL: NCT00767026
Title: COPE Intervention for Parents of Children With Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Lisa V. Duffy PhD(c), CPNP-PC, CNRN, Children's Hospital Boston
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1F31NR010645-01 (NIH); F31NR010645 (NIH)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Caregiver Burden; Parenting a Child with a Chronic Illness
MeSH Terms: conditions — Epilepsy; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: COPE (Creating Opportunities for Parent Empowerment)
- 2 (Active Comparator)
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: COPE (Creating Opportunities for Parent Empowerment) — Twenty-four hours after admission to the hospital, this group will receive Phase I of the study which includes information focusing on what parents can expect during their child's hospital stay, and how they can help their child cope with the experience. Prior to discharge parents will receive additional information pertaining to Phase II of the study. At 3 days post discharge, the participants will receive a follow up phone call to reiterate the information provided in Phase II and ask parents about questions or problems since discharge. One week following, participants will be asked to complete assessments. At 6 weeks after the hospitalization they will receive Phase III, which includes, additional information on behaviors parents can expect to see in their children following a hospitalization. Parents will be given a workbook that will teach them techniques to help their child cope. Then at 6 weeks after the last intervention phase, participants will again complete assessments.
  Arms: 1
Behavioral: Standard education — This group will receive standard education regarding medication management and seizure first aid. This group will also receive information, oral and written, that will discuss tests to be administered during the hospitalization. The usual care group also receives a call at home within one week after discharge from a nurse to ask if they had any problems with their stay, and if they have any further needs or questions.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the program Creating Opportunities for Parent Empowerment (COPE) is feasible to administer to parents of children with neurological conditions. The goal of the study is to empower parents by providing them with educational materials designed to teach them how to foster healthy coping skills in their child.

DETAILED DESCRIPTION:
Chronic neurological conditions have a significant impact on the child and family system. Parents of children with neurological conditions want to foster the healthy development of their child, however, they struggle with constant feelings of uncertainty, which results in an increased level of stress that can interfere with this goal. Stress in parents also results in anxiety, depression, decreased confidence in care giving skills, ultimately leading to an increase in behavior problems in the child with epilepsy. Pediatric nurses are in a position to intervene with parents of children with epilepsy to facilitate coping with and adjustment to these issues.

Although many researchers have identified the relationship between effective parental coping and the improved psychosocial outcomes of children with epilepsy, little has been done to test interventions that may be effective in improving the coping strategies of parents of children with epilepsy. COPE (Creating Opportunities for Parent Empowerment) is a nurse coached educational intervention, which shows promise for improving coping in parents of hospitalized children. This is particularly significant for parents of children with neurological conditions, as these conditions are associated with repeated hospitalizations, stigma, and numerous comorbidities. Collectively, these factors make epilepsy one of the most stress producing pediatric conditions for parents to manage.

This study will help to advance Nursing science in several ways. First, this study will develop an intervention that can be used to teach parents how to help their children cope with living with a chronic condition. This intervention could further advance Nursing science because it could be adapted and trials performed with children who have a wide variety of medical conditions. This study has the potential to improve the way we prepare parents and children for hospitalization. This study will guide nursing in how to best help families cope with caring for a child with a chronic condition.

The research consent form has been reviewed and approved by the IRB at both Children's Hospital Boston and Boston College. The consent form addresses the following topics:

A. Why the research is being conducted and what is its purpose B. Who is conducting the study and where it is being conducted C. How individuals are selected to be in the study and how many will participate D. What the participant needs to do in the research study E. What are the risks of the study and what could go wrong F. What are the benefits of the study G. Costs and payments associated with the study H. What happens to the information obtained from the study and what about confidentiality I. What are the choices if the participant does not want to be involved with the study J. What are the rights of a research participant K. HIPAA

ELIGIBILITY:
Inclusion Criteria:

* Parents of children ages 2-6 with epilepsy
* Children must have been diagnosed with epilepsy for a minimum period of six months
* Parents of children currently admitted to the Children's Hospital Boston inpatient neuroscience unit (CHB-INU) for long term EEG
* High school graduate literate in English
* Access to cellular or home telephone

Exclusion Criteria:

* Parents of children who have been diagnosed with co-morbid conditions including, but not limited to: cancer, mitochondrial or metabolic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Parental depression | 24 hours, 1-, 8 -, and 12- weeks after discharge
Parental Anxiety | 24 hours, 1-, 8 -, and 12- weeks after discharge
Confidence in Parenting Skills | 24 hours, 1-, 8 -, and 12- weeks after discharge

SECONDARY OUTCOMES:
Behavior problems in the child | 24 hours, 1-, 8 -, and 12- weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lisa V Duffy, PhD(c), CPNP-PC, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Amdam, A., Langslet, B., & Holmseth, T. (2001). The penguin: A teaching Ppan for children with epilepsy. In: Pfafflin, M., Fraser, Thorbecke et al. (Eds). Comprehensive care for people with epilepsy. London: John Libbey.
- [Background] Austin JK, Dunn DW. Children with epilepsy: quality of life and psychosocial needs. Annu Rev Nurs Res. 2000;18:26-47. PMID 10918931
- [Background] Austin JK, Harezlak J, Dunn DW, Huster GA, Rose DF, Ambrosius WT. Behavior problems in children before first recognized seizures. Pediatrics. 2001 Jan;107(1):115-22. doi: 10.1542/peds.107.1.115. PMID 11134444
- [Background] Austin, J.K., McNelis, A.M., Shore, C.P., Dunn, D.W., & Musick, B. (2002). A feasibility study of a family seizure management program: "Be Seizure Smart." Journal of Neuroscience Nursing, 34(1), 30-37.
- [Background] Austin JK, Dunn DW, Johnson CS, Perkins SM. Behavioral issues involving children and adolescents with epilepsy and the impact of their families: recent research data. Epilepsy Behav. 2004 Oct;5 Suppl 3:S33-41. doi: 10.1016/j.yebeh.2004.06.014. PMID 15351344
- [Background] Aytch LS, Hammond R, White C. Seizures in infants and young children: an exploratory study of family experiences and needs for information and support. J Neurosci Nurs. 2001 Oct;33(5):278-85. doi: 10.1097/01376517-200110000-00008. PMID 11668886
- [Background] Bazil CW. Comprehensive care of the epilepsy patient--control, comorbidity, and cost. Epilepsia. 2004;45 Suppl 6:3-12. doi: 10.1111/j.0013-9580.2004.455002.x. PMID 15315510
- [Background] Berg AT, Smith SN, Frobish D, Levy SR, Testa FM, Beckerman B, Shinnar S. Special education needs of children with newly diagnosed epilepsy. Dev Med Child Neurol. 2005 Nov;47(11):749-53. doi: 10.1017/S001216220500157X. PMID 16225738
- [Background] Buelow JM, McNelis A, Shore CP, Austin JK. Stressors of parents of children with epilepsy and intellectual disability. J Neurosci Nurs. 2006 Jun;38(3):147-54, 176. doi: 10.1097/01376517-200606000-00003. PMID 16817666
- [Background] Carlton-Ford S, Miller R, Nealeigh N, Sanchez N. The effects of perceived stigma and psychological over-control on the behavioural problems of children with epilepsy. Seizure. 1997 Oct;6(5):383-91. doi: 10.1016/s1059-1311(97)80038-6. PMID 9663802
- [Background] Chapieski L, Brewer V, Evankovich K, Culhane-Shelburne K, Zelman K, Alexander A. Adaptive functioning in children with seizures: impact of maternal anxiety about epilepsy. Epilepsy Behav. 2005 Sep;7(2):246-52. doi: 10.1016/j.yebeh.2005.05.002. PMID 15996525
- [Background] Hufford, B.S., Glueckauf, R.L., & Webb, P.M. (1999). Home-based, interactive videoconferencing for adolescents with epilepsy and their families. Rehabilitation Psychology, 44(2), 176-193.
- [Background] Jacoby A, Snape D, Baker GA. Epilepsy and social identity: the stigma of a chronic neurological disorder. Lancet Neurol. 2005 Mar;4(3):171-8. doi: 10.1016/S1474-4422(05)01014-8. PMID 15721827
- [Background] Keller D, Honig AS. Maternal and paternal stress in families with school-aged children with disabilities. Am J Orthopsychiatry. 2004 Jul;74(3):337-48. doi: 10.1037/0002-9432.74.3.337. PMID 15291710
- [Background] Low SM, Stocker C. Family functioning and children's adjustment: associations among parents' depressed mood, marital hostility, parent-child hostility, and children's adjustment. J Fam Psychol. 2005 Sep;19(3):394-403. doi: 10.1037/0893-3200.19.3.394. PMID 16221020
- [Background] Melnyk BM. Coping with unplanned childhood hospitalization: effects of informational interventions on mothers and children. Nurs Res. 1994 Jan-Feb;43(1):50-5. PMID 8295841
- [Background] Melnyk BM. Parental coping with childhood hospitalization: a theoretical framework to guide research and clinical interventions. Matern Child Nurs J. 1995 Oct-Dec;23(4):123-31. PMID 8826078
- [Background] Melnyk BM, Alpert-Gillis LJ, Hensel PB, Cable-Beiling RC, Rubenstein JS. Helping mothers cope with a critically ill child: a pilot test of the COPE intervention. Res Nurs Health. 1997 Feb;20(1):3-14. doi: 10.1002/(sici)1098-240x(199702)20:13.0.co;2-q. PMID 9024473
- [Background] Melnyk BM, Alpert-Gillis LJ. The COPE program: a strategy to improve outcomes of critically ill young children and their parents. Pediatr Nurs. 1998 Nov-Dec;24(6):521-7. PMID 10085993
- [Background] Melnyk BM, Feinstein NF, Moldenhouer Z, Small L. Coping in parents of children who are chronically ill: strategies for assessment and intervention. Pediatr Nurs. 2001 Nov-Dec;27(6):548-58. PMID 12024526
- [Background] Melnyk BM, Alpert-Gillis L, Feinstein NF, Crean HF, Johnson J, Fairbanks E, Small L, Rubenstein J, Slota M, Corbo-Richert B. Creating opportunities for parent empowerment: program effects on the mental health/coping outcomes of critically ill young children and their mothers. Pediatrics. 2004 Jun;113(6):e597-607. doi: 10.1542/peds.113.6.e597. PMID 15173543
- [Background] Mu PF, Wong TT, Chang KP, Kwan SY. Predictors of maternal depression for families having a child with epilepsy. J Nurs Res. 2001 Sep;9(4):116-26. PMID 11789131
- [Background] Mu PF. Paternal reactions to a child with epilepsy: uncertainty, coping strategies, and depression. J Adv Nurs. 2005 Feb;49(4):367-76. doi: 10.1111/j.1365-2648.2004.03300.x. PMID 15701151
- [Background] Mu PF, Kuo HC, Chang KP. Boundary ambiguity, coping patterns and depression in mothers caring for children with epilepsy in Taiwan. Int J Nurs Stud. 2005 Mar;42(3):273-82. doi: 10.1016/j.ijnurstu.2004.07.002. PMID 15708014
- [Background] Oostrom KJ, Schouten A, Kruitwagen CL, Peters AC, Jennekens-Schinkel A; Dutch Study Group of Epilepsy in Childhood. Parents' perceptions of adversity introduced by upheaval and uncertainty at the onset of childhood epilepsy. Epilepsia. 2001 Nov;42(11):1452-60. doi: 10.1046/j.1528-1157.2001.14201.x. PMID 11879349
- [Background] Sawin KJ, Lannon SL, Austin JK. Camp experiences and attitudes toward epilepsy: a pilot study. J Neurosci Nurs. 2001 Feb;33(1):57-64. doi: 10.1097/01376517-200102000-00008. PMID 11233363
- [Background] Shore CP, Austin JK, Huster GA, Dunn DW. Identifying risk factors for maternal depression in families of adolescents with epilepsy. J Spec Pediatr Nurs. 2002 Apr-Jun;7(2):71-80. doi: 10.1111/j.1744-6155.2002.tb00153.x. PMID 12061495
- [Background] Snead K, Ackerson J, Bailey K, Schmitt MM, Madan-Swain A, Martin RC. Taking charge of epilepsy: the development of a structured psychoeducational group intervention for adolescents with epilepsy and their parents. Epilepsy Behav. 2004 Aug;5(4):547-56. doi: 10.1016/j.yebeh.2004.04.012. PMID 15256193
- [Background] Tieffenberg JA, Wood EI, Alonso A, Tossutti MS, Vicente MF. A randomized field trial of ACINDES: a child-centered training model for children with chronic illnesses (asthma and epilepsy). J Urban Health. 2000 Jun;77(2):280-97. doi: 10.1007/BF02390539. PMID 10856009
- [Background] Thomas SV, Bindu VB. Psychosocial and economic problems of parents of children with epilepsy. Seizure. 1999 Feb;8(1):66-9. doi: 10.1053/seiz.1998.0241. PMID 10091852
- [Background] Williams J, Steel C, Sharp GB, DelosReyes E, Phillips T, Bates S, Lange B, Griebel ML. Parental anxiety and quality of life in children with epilepsy. Epilepsy Behav. 2003 Oct;4(5):483-6. doi: 10.1016/s1525-5050(03)00159-8. PMID 14527488